CLINICAL TRIAL: NCT01714245
Title: A Multicenter, Prospective Study to Evaluate CLn® BodyWash As An Adjunctive Therapy in Pediatric Subjects With Moderate to Severe, Staphylococcus Aureus Colonized Atopic Dermatitis
Brief Title: A Study to Evaluate CLn® BodyWash As Added Therapy in Eczema Patients
Acronym: CLeaN
Status: Completed | Type: Observational
Sponsor: TopMD Skin Care, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN 003.6
Record Dates: First submitted 2012-10-18; First posted 2012-10-25 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Eczema; Atopic Dermatitis
Keywords: Eczema; Atopic Dermatitis; Compromised Skin; Inflamed Skin
MeSH Terms: conditions — Eczema; Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if CLn BodyWash, a novel new gel cleanser formulated with surfactants and preserved with sodium hypochlorite, is effective at decreasing severity, body surface area and itching for patients with Atopic Dermatitis, or eczema.

DETAILED DESCRIPTION:
Staphylococcus aureus colonization and potential infection represent a common clinical finding in patients with atopic dermatitis (AD) and may contribute to exacerbation of the disease. Atopic patients are commonly colonized with S. aureus on both lesional and non-lesional skin. Antibiotic treatment of clinically infected patients can often improve the bacterial infection as well as reduce the overall severity of AD. More recently, measures to reduce S. aureus colonization have been shown to decrease the clinical severity of Atopic Dermatitis in patients with clinical signs of secondary bacterial infection of the skin.

Given the increasing incidence of recurrent skin infections caused by S. aureus, measures such as dilute sodium hypochlorite (bleach) baths have been adopted by many physicians in an effort to decrease infection rates and disease severity in patients with atopic dermatitis, recurrent impetigo, cellulitis, folliculitis, boils and abscesses. There is some controversy in the literature regarding the efficacy of anti-staphylococcal treatments in improving AD in patients without active clinical infection as one review noted limited benefit while another study showed that dilute bleach baths improved AD.

Bleach baths are widely used in pediatrics and adult medicine. A common regimen consists of adding ½ cup of household bleach into ½ tub of warm bath water, resulting in a 0.009% sodium hypochlorite concentration. (www.bleachbath.com) CLn® BodyWash contains several common surfactants to clean the skin and 0.006% sodium hypochlorite concentration for preservation, and is further diluted when lathered onto the skin with water. This over the counter product is delivered in a sealed, easy to use dispenser, which can be used in the bath or shower, lathered on and rinsed off after 1-2 minutes of skin contact. CLn® BodyWash may be a convenient alternative to bleach baths.

ELIGIBILITY:
Inclusion Criteria:

* 6 months to 18 years
* moderate to severe Atopic Dermatitis
* positive staphylococcus aureus skin culture

Exclusion Criteria:

* active clinical infection
* on antibiotics in the last 4 weeks
* on immunosuppression drug in the last 4 weeks
* using bleach bath in the last 2 weeks
* able to maintain current regimen

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with Atopic Dermatitis
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Improvement in Health of Skin EASI | 6 weeks
  Change from baseline in Eczema Area Severity Index (EASI) Score.
Improvement in Health of Skin IGA | 6 weeks
  Change from baseline in Investigator Global Assessment (IGA) Score.
Improvement in Health of Skin BSA | 6 weeks
  Change from baseline in Body Surface Area (BSA) Score.

SECONDARY OUTCOMES:
Patient satisfaction | 6 weeks
  Quality of Life Questionnaires will be reviewed for a patient and family satisfaction.
Decreased itching | 6 weeks
  Visual Analog Scale will be reviewed for decrease in pruritus.
Reduction of bacteria | 6 weeks
  Bacterial cultures will be evaluated for decreased quantitative numbers.

CONTACTS AND LOCATIONS:
Overall Officials: Adelaide A. Hebert, MD, Principal Investigator — University of Texas Medical School - Houston
Locations (2):
- United States (2):
  - Northwestern University, Department of Dermatology, Chicago, Illinois
  - University of Texas Medical School - Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Majewski S, Bhattacharya T, Asztalos M, Bohaty B, Durham KC, West DP, Hebert AA, Paller AS. Sodium hypochlorite body wash in the management of Staphylococcus aureus-colonized moderate-to-severe atopic dermatitis in infants, children, and adolescents. Pediatr Dermatol. 2019 Jul;36(4):442-447. doi: 10.1111/pde.13842. Epub 2019 Apr 15. PMID 30983053